CLINICAL TRIAL: NCT03786471
Title: Comparative Effectiveness of Health System-based Versus Community-Based Dementia Care / A Pragmatic Clinical Trial of the Effectiveness and Cost-Effectiveness of Dementia Care
Brief Title: D-CARE - The Dementia Care Study: A Pragmatic Clinical Trial of Health System-Based Versus Community-Based Dementia Care
Acronym: D-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Institute on Aging (NIA) (NIH); Yale University (Other); Benjamin Rose Institute on Aging (Other); Baylor Scott and White Health (Other); Wake Forest University Health Sciences (Other); University of Texas (Other); Geisinger Clinic (Other); University of Oklahoma (Other); RAND (Other)
Responsible Party: Principal Investigator, David B. Reuben, MD, Director, Multicampus Program in Geriatric Medicine & Gerontology; Chief, Division of Geriatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB 18-001796; R01AG061078-01 (NIH); PCS-2017C1-6534 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2018-12-17; First posted 2018-12-26 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Dementia
Keywords: dementia; pragmatic clinical trial; effectiveness; cost-effectiveness; Alzheimer's disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: * 2150 dyads of persons with dementia and their respective primary caregiver
  * 1000 in each intervention arm, and 150 in the usual care arm
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Systems-Based Dementia Care (Active Comparator): Dementia care that is based in the health care system, which partners with community-based organizations to provide comprehensive, coordinated, patient-centered care. The health system-based dementia care arm uses a Dementia Care Specialist (Nurse Practitioner or Physician Assistant) supervised by a physician to tailor and facilitate dementia care delivery in collaboration with the primary care physician (co-management). The Health Systems-Based Dementia Care arm is based on UCLA's Alzheimer's and Dementia Care Program.
  Interventions: Other: Health System-based Dementia Care
- Community-Based Dementia Care (Active Comparator): Dementia care that is based in community organizations, which gives equal attention to patients and their primary family or friend caregivers. The community-based dementia care arm uses Care Consultants (social workers, nurses, or licensed therapist). Patients with dementia are engaged in the program whenever possible. Caregivers can be the sole program participant, when patients are too impaired. The program establishes a long-term relationship between Care Consultants and families. The exact content of assistance provided is tailored to the preferences of individual patients and caregivers, and is holistic in the range of potential concerns of problems addressed. The Community-Based Dementia Care arm is based on the Benjamin Rose Institute on Aging's Care Consultation Program.
  Interventions: Other: Community-based Dementia Care
- Usual Care (Other): Dementia care that most closely corresponds to traditional care. This arm will also receive standardized educational materials (hard copies and internet-based resources), referral to the Alzheimer's Association 1-800 national helpline to speak to a master's level consultant for decision-making support, crisis assistance, and caregiver education, as well as referral to local programs and services.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Health System-based Dementia Care — Active comparator
  Arms: Health Systems-Based Dementia Care
Other: Community-based Dementia Care — Active comparator
  Arms: Community-Based Dementia Care
Other: Usual Care — Control
  Arms: Usual Care

SUMMARY:
D-CARE: The Dementia Care Study

This pragmatic randomized clinical trial of 2150 persons with dementia and their caregivers, at four diverse clinical trial sites in the United States, compares the effectiveness and cost-effectiveness of 18 months of health systems-based dementia care provided by a Dementia Care Specialist (nurse practitioner or physician assistant) who works within the heath system versus community-based dementia care provided by a Care Consultant (social worker, nurse, or therapist) who works at a Community-Based Organization (CBO).

The trial will also compare the effectiveness and cost-effectiveness of both models versus usual care.

DETAILED DESCRIPTION:
D-CARE: The Dementia Care Study

Objective: To determine the comparative effectiveness and cost-effectiveness of two evidence-based models of comprehensive dementia care, as well as the effectiveness and cost-effectiveness of both models versus usual care.

Design: A pragmatic randomized 3-arm superiority trial. The unit of randomization is the patient/caregiver dyad.

Duration: 6.5 years. This includes 34 months for recruitment of study participants, 18 months of interventions/usual care, and simultaneously 18 months of follow-up for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* The person with dementia has a diagnosis of dementia established by a physician or other primary care provider
* The person with dementia has a primary care provider who is willing to partner with the study
* The person with dementia has a caregiver who speaks English or Spanish, and has a phone
* Persons living with dementia in assisted living facilities will be eligible if they do not meet any exclusion criteria (however, no more than 25% of participants can be living in assisted living facilities at the time of enrollment. This will be monitored when the first 25% of the sample has been enrolled.)

Exclusion Criteria:

* The person with dementia resides in a nursing home at the time of recruitment
* The person with dementia is enrolled in hospice at the time of screen
* The person with dementia plans to move out of the area within the coming year
* The caregiver of the person with dementia is unwilling or anticipates being incapable of providing self-reported outcome measures for 18 months
* Baseline measures refused or not completed
* The caregiver is paid, and is not a relative or close friend of the person with dementia
* At telephone or in-person screener, the caregiver has cognitive impairment
* The person with dementia or caregiver is participating in another dementia intervention study
* Patients and caregivers who are members of a sites' Local Patient & Stakeholder Committee
* There is already a member of the same household participating in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2176 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reuben, MD, Principal Investigator — University of California, Los Angeles; Thomas Gill, MD, Principal Investigator — Yale University; David Bass, PhD, Principal Investigator — Benjamin Rose Institute on Aging; Lee Jennings, MD, Principal Investigator — University of Oklohoma; Maya Lichtenstein, MD, Principal Investigator — Geisinger Clinic; Peter Peduzzi, PhD, Principal Investigator — Yale University; Alan Stevens, PhD, Principal Investigator — Baylor Scott and White Health; Elena Volpi, MD, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Jeffrey Williamson, MD, Principal Investigator — Wake Forest University Health Sciences; Christopher Callahan, MD, Study Chair — Indiana University; Katie Maslow, MSW, Study Chair — Gerontological Society of America; Jenny Summapund, MA, Study Director — University of California, Los Angeles
Locations (4):
- United States (4):
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Geisinger Health, Wilkes-Barre, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor Scott & White, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oyeyemi DM, Greene EJ, Xu Y, Lee DR, Samper-Ternent R, Lichtenstein ML, Stevens A, Williamson JD, Karlamangla AS, Saliba D, Reuben DB. Self-efficacy change among diverse family caregivers in dementia care. J Gerontol B Psychol Sci Soc Sci. 2026 Jan 12;81(2):gbaf233. doi: 10.1093/geronb/gbaf233. PMID 41243731
- [Derived] Reuben DB, Stevens AB, Gill TM, Williamson J, Volpi E, Lichtenstein ML, Jennings LA, Galloway R, Summapund J, Araujo K, Bass D, Weitzman L, Tan ZS, Evertson LC, Yang M, Green AS, Samper-Ternent R, Borek P, Xu Y, Peduzzi P, Greene EJ; D-CARE Study. Patient and Caregiver Outcomes of Health System, Community-Based, and Usual Dementia Care: A Prespecified Analysis of the Dementia Care Study (D-CARE) Randomized Clinical Trial. JAMA Intern Med. 2025 Oct 1;185(10):1227-1236. doi: 10.1001/jamainternmed.2025.4247. PMID 40892399
- [Derived] Reuben DB, Gill TM, Stevens A, Williamson J, Volpi E, Lichtenstein M, Jennings LA, Galloway R, Summapund J, Araujo K, Bass D, Weitzman L, Tan ZS, Evertson L, Yang M, Currie K, Green AS, Godoy S, Abraham S, Reese J, Samper-Ternent R, Hirst RM, Borek P, Charpentier P, Meng C, Dziura J, Xu Y, Skokos EA, He Z, Aiudi S, Peduzzi P, Greene EJ; D-CARE Study. Health System, Community-Based, or Usual Dementia Care for Persons With Dementia and Caregivers: The D-CARE Randomized Clinical Trial. JAMA. 2025 Mar 18;333(11):950-961. doi: 10.1001/jama.2024.25056. PMID 39878968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred by physicians or self-referred at 4 clinical trial sites (2 academic, 2 community-based) in 3 states. 2,176 PLwD/caregiver dyads were enrolled between June 2019 and January 2022.
Pre-assignment Details: Of 11,652 referred for screening, 156 were not screened due to recruitment ending, 2,929 could not be screened, 290 were unable to complete the baseline interview, 3,415 met exclusion criteria, and 2,686 declined participation.
Groups:
- Usual Care: Dementia care that most closely corresponds to traditional care. This arm will also receive standardized educational materials (hard copies and internet-based resources), referral to the Alzheimer's Association 1-800-3900 national helpline to speak to a master's level consultant for decision-making support, crisis assistance, and caregiver education, as well as referral to local programs and services.
  Usual Care: Control
Period: Overall Study
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Started | 1016 | 1016 | 144
Completed 3-month Interview | 830 | 872 | 120
Completed 6-month Interview | 804 | 821 | 112
Completed 12-month Interview | 702 | 733 | 93
Completed | 600 | 662 | 81
Not Completed | 416 | 354 | 63
Not completed — Death | 254 | 223 | 37
Not completed — Lost to Follow-up | 63 | 50 | 15
Not completed — Withdrawal by Subject | 99 | 81 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care | Total
Number analyzed (Participants) | 1016 | 1016 | 144 | 2176
Age, Continuous [Mean (Standard Deviation); unit: years]
  Caregiver Age | 64.8 (12.3) | 65.6 (12.3) | 66.2 (11.7) | 65.2 (12.3)
  PLWD Age | 80.6 (8.3) | 80.6 (8.7) | 81.0 (8.4) | 80.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  PLWD Sex: Female | 611 | 583 | 77 | 1271
  PLWD Sex: Male | 405 | 433 | 67 | 905
  Caregiver Sex: Female | 772 | 760 | 118 | 1650
  Caregiver Sex: Male | 244 | 256 | 26 | 526
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of persons living with dementia (PLWD)
  Participants
    Hispanic or Latino | 90 | 87 | 14 | 191
    Not Hispanic or Latino | 925 | 928 | 130 | 1983
    Unknown or Not Reported | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of caregivers
  Participants
    Hispanic or Latino | 95 | 94 | 16 | 205
    Not Hispanic or Latino | 919 | 922 | 128 | 1969
    Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of caregivers
  Participants
    American Indian or Alaska Native | 4 | 4 | 0 | 8
    Asian | 8 | 3 | 0 | 11
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 121 | 113 | 18 | 252
    White | 855 | 872 | 119 | 1846
    More than one race | 10 | 11 | 2 | 23
    Unknown or Not Reported | 18 | 13 | 5 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of persons living with dementia (PLWD)
  Participants
    American Indian or Alaska Native | 4 | 4 | 1 | 9
    Asian | 10 | 3 | 0 | 13
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 124 | 115 | 20 | 259
    White | 847 | 873 | 119 | 1839
    More than one race | 7 | 5 | 1 | 13
    Unknown or Not Reported | 24 | 16 | 3 | 43
Region of Enrollment [Number; unit: dyads]
  United States | 1016 | 1016 | 144 | 2176
Caregiver Education [Count of Participants; unit: Participants]
  Less than HS graduate | 39 | 28 | 1 | 68
  HS graduate or GED | 172 | 164 | 22 | 358
  Some college or equivalent | 303 | 301 | 43 | 647
  Graduated from college | 302 | 327 | 46 | 675
  Graduate or professional degree | 200 | 196 | 32 | 428
  Unknown or not reported | 0 | 0 | 0 | 0
PLWD Education [Count of Participants; unit: Participants]
  Less than HS graduate | 167 | 154 | 18 | 339
  HS graduate or GED | 267 | 312 | 48 | 627
  Some college or equivalent | 238 | 238 | 35 | 511
  Graduated from college | 206 | 168 | 21 | 395
  Graduate or professional degree | 136 | 144 | 20 | 300
  Unknown or not reported | 2 | 0 | 2 | 4
Caregiver Primary Language [Count of Participants; unit: Participants]
  English | 1011 | 1004 | 144 | 2159
  Spanish | 5 | 12 | 0 | 17
Persons Living with Dementia (PLWD) Primary Language [Count of Participants; unit: Participants]
  English | 999 | 995 | 142 | 2136
  Spanish | 17 | 21 | 2 | 40
Caregiver Marital Status [Count of Participants; unit: Participants]
  Married/Partner | 780 | 799 | 118 | 1697
  Widowed | 25 | 27 | 1 | 53
  Divorced | 97 | 98 | 13 | 208
  Single | 105 | 84 | 9 | 198
  Other | 9 | 8 | 3 | 20
PLWD Marital Status [Count of Participants; unit: Participants]
  Married/Partner | 547 | 546 | 78 | 1171
  Widowed | 322 | 346 | 51 | 719
  Divorced | 99 | 97 | 12 | 208
  Single | 40 | 22 | 3 | 65
  Other | 8 | 5 | 0 | 13
Caregiver living with PLWD [Count of Participants; unit: Participants]
  Yes | 728 | 755 | 105 | 1588
  No | 287 | 261 | 39 | 587
  Unknown or not reported | 1 | 0 | 0 | 1
PLWD Living Arrangement [Count of Participants; unit: Participants]
  At home alone without caregiver | 139 | 130 | 21 | 290
  At home with caregiver | 723 | 753 | 105 | 1581
  At home with someone else | 97 | 83 | 9 | 189
  Assisted Living Facility | 57 | 50 | 9 | 116

OUTCOME MEASURES:

1. Primary Outcome: Severity of Dementia-related Behavioral Symptoms
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 992 | 990 | 140
score on a scale | 10.32 (0.22) | 9.93 (0.21) | 10.42 (0.56)

2. Primary Outcome: Severity of Dementia-related Behavioral Symptoms
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 3 month.
Time Frame: 3-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 776 | 831 | 114
score on a scale | 9.10 (0.24) | 8.98 (0.22) | 9.67 (0.65)

3. Primary Outcome: Severity of Dementia-related Behavioral Symptoms
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 6 months.
Time Frame: 6-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 764 | 784 | 107
score on a scale | 9.41 (.25) | 8.78 (.23) | 9.93 (.68)

4. Primary Outcome: Severity of Dementia-related Behavioral Symptoms
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 12 months.
Time Frame: 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 665 | 685 | 87
score on a scale | 9.58 (.27) | 9.14 (.25) | 9.95 (.74)

5. Primary Outcome: Severity of Dementia-related Behavioral Symptoms
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 18 months.
Time Frame: 18-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 564 | 620 | 75
score on a scale | 9.80 (0.29) | 9.51 (0.27) | 9.60 (0.79)

6. Primary Outcome: Severity of Dementia-related Behavioral Symptoms (Common Baseline)
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the least squares mean of the baseline "treatment 0", which can be compared to the overall follow-up least square means to estimate treatment effects in each arm.
Time Frame: Baseline
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Groups:
- Common Baseline: Constrained Longitudinal Model. All groups are assigned a common "treatment 0" at baseline.
Arm/Group | Common Baseline
Number analyzed (Participants) | 2166
score on a scale | 10.07 [9.71 to 10.43]

7. Primary Outcome: Severity of Dementia-related Behavioral Symptoms
Description: The severity of symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Severity (NPI-Q Severity). The NPI-Q Severity is a validated survey that assesses the caregiver's perception of the severity of 12 dementia-related psychiatric and behavioral symptoms. NPI-Q Severity score ranges from 0-36 with higher scores indicating more severe symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents those average least squares means across all follow-up times for each arm.
Time Frame: Average of 3M, 6M, 12M, and 18M least square means.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1012 | 1011 | 143
score on a scale | 9.79 [9.37 to 10.22] | 9.50 [9.08 to 9.91] | 10.12 [9.15 to 11.08]
Statistical Analysis 1: Comparison: Health Systems-Based Dementia Care vs Community-Based Dementia Care; Test type: Superiority; p = 0.33, Mixed Models Analysis — Alpha = 0.025; Hochberg correction for three pairwise comparisons; marginal difference of LS means = 0.30, 97.5% CI 2-sided [-0.18 to 0.78]
Statistical Analysis 2: Comparison: Community-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.33, Mixed Models Analysis — Alpha = 0.025; Hochberg correction for three pairwise comparisons; marginal difference of LS means = -0.62, 97.5% CI 2-sided [-1.61 to 0.37]
Statistical Analysis 3: Comparison: Health Systems-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.46, Mixed Models Analysis — Alpha = 0.025; Hochberg correction for three pairwise comparisons; marginal difference of LS means = -0.33, 97.5% CI 2-sided [-1.32 to 0.67]

8. Primary Outcome: Caregiver Distress/Strain
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1004 | 1007 | 141
score on a scale | 11.03 (0.20) | 10.65 (0.19) | 11.13 (0.55)

9. Primary Outcome: Caregiver Distress/Strain
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 3 months.
Time Frame: 3-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 820 | 855 | 120
score on a scale | 10.52 (0.22) | 10.01 (0.20) | 10.00 (0.53)

10. Primary Outcome: Caregiver Distress/Strain
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 6 months.
Time Frame: 6-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 790 | 809 | 112
score on a scale | 10.61 (0.23) | 10.26 (0.22) | 10.53 (0.65)

11. Primary Outcome: Caregiver Distress/Strain
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 12 months.
Time Frame: 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 685 | 716 | 92
score on a scale | 11.00 (0.24) | 10.50 (0.24) | 10.41 (0.69)

12. Primary Outcome: Caregiver Distress/Strain
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 18 months.
Time Frame: 18-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 584 | 646 | 79
score on a scale | 11.26 (0.26) | 10.64 (0.24) | 10.32 (0.72)

13. Primary Outcome: Caregiver Distress/Strain (Common Baseline)
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the least squares mean of the baseline "treatment 0", which can be compared to the overall follow-up least square means to estimate treatment effects in each arm.
Time Frame: Baseline
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Common Baseline
Number analyzed (Participants) | 2171
score on a scale | 10.61 [10.29 to 10.93]

14. Primary Outcome: Caregiver Distress/Strain
Description: The level of caregiver distress/strain as measured by the Modified Caregiver Strain Index (MCSI). The MCSI is a 13-item validated tool used to assess severity of caregiver strain. The index targets financial, physical, psychological, and social aspects of strain and is scored from 0 to 26 with higher scores indicating greater levels of strain. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents those average least squares means across all follow-up times for each arm.
Time Frame: Average of 3M, 6M, 12M, and 18M least square means
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1013 | 1014 | 144
score on a scale | 10.74 [10.36 to 11.12] | 10.50 [10.12 to 10.87] | 10.60 [9.77 to 11.42]
Statistical Analysis 1: Comparison: Health Systems-Based Dementia Care vs Community-Based Dementia Care; Test type: Superiority; p = 0.54, Mixed Models Analysis — Alpha = 0.025; Hochberg correction for three pairwise comparisons; marginal difference of LS means = 0.25, 97.5% CI 2-sided [-0.16 to 0.66]
Statistical Analysis 2: Comparison: Community-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.79, Mixed Models Analysis — Alpha = 0.025; Hochberg correction for three pairwise comparisons; marginal difference of LS means = -0.10, 97.5% CI 2-sided [-0.94 to 0.74]
Statistical Analysis 3: Comparison: Health Systems-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.79, Mixed Models Analysis — Alpha = 0.025; Hochberg correction for three pairwise comparisons; marginal difference of LS means = 0.14, 97.5% CI 2-sided [-0.70 to 0.99]

15. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 996 | 991 | 141
score on a scale | 12.96 (0.32) | 12.66 (0.31) | 12.69 (0.79)

16. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 3 months.
Time Frame: 3-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 793 | 834 | 114
score on a scale | 11.45 (0.35) | 11.15 (0.32) | 12.42 (0.91)

17. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 6 months.
Time Frame: 6-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 763 | 785 | 106
score on a scale | 11.88 (0.37) | 11.23 (0.34) | 12.62 (0.95)

18. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 12 months.
Time Frame: 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 666 | 686 | 86
score on a scale | 12.09 (0.39) | 11.76 (0.37) | 12.63 (1.02)

19. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 18 months.
Time Frame: 18-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 564 | 622 | 75
score on a scale | 12.12 (0.43) | 11.80 (0.40) | 11.53 (1.12)

20. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms (Common Baseline)
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the least squares mean of the baseline "treatment 0", which can be compared to the overall follow-up least square means to estimate treatment effects in each arm.
Time Frame: Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Common Baseline
Number analyzed (Participants) | 2166
score on a scale | 12.62 [12.16 to 13.08]

21. Secondary Outcome: Level of Distress Experienced by the Caregiver in Response to Dementia-related Psychiatric and Behavioral Symptoms
Description: Distress of caregivers due to the symptoms of psychopathology in persons with dementia as measured by the Neuro-Psychiatric Inventory Questionnaire - Distress (NPI-Q Distress). The NPI-Q Distress scale is a validated survey that assesses the level of distress experienced by the caregiver in response to dementia-related psychiatric and behavioral symptoms. NPI-Q Distress score ranges from 0-60 with higher scores indicating more severe distress. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents those average least squares means across all follow-up times for each arm.
Time Frame: Average of 3M, 6M, 12M, and 18M least square means
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1013 | 1010 | 143
score on a scale | 12.29 [11.76 to 12.83] | 11.77 [11.25 to 12.30] | 13.10 [11.88 to 14.32]
Statistical Analysis 1: Comparison: Health Systems-Based Dementia Care vs Community-Based Dementia Care; Test type: Superiority; p = 0.48, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = 0.52, 95% CI 2-sided [-.09 to 1.13]
Statistical Analysis 2: Comparison: Health Systems-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.62, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons *three secondary outcomes; marginal difference of LS means = -.81, 95% CI 2-sided [-2.07 to 0.45]
Statistical Analysis 3: Comparison: Community-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.23, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = -1.33, 95% CI 2-sided [-2.58 to -0.07]

22. Secondary Outcome: Severity of Depression in Caregivers
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1009 | 1009 | 144
score on a scale | 4.72 (0.15) | 4.78 (0.15) | 5.17 (.40)

23. Secondary Outcome: Severity of Depression in Caregivers
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 3 months.
Time Frame: 3-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 825 | 866 | 120
score on a scale | 4.47 (0.16) | 4.40 (.15) | 4.68 (.41)

24. Secondary Outcome: Severity of Depression in Caregivers
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 6 months.
Time Frame: 6-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 788 | 813 | 112
score on a scale | 4.55 (.16) | 4.26 (.15) | 4.57 (.42)

25. Secondary Outcome: Severity of Depression in Caregivers
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 12 months.
Time Frame: 12-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 685 | 719 | 92
score on a scale | 4.46 (.17) | 4.41 (.17) | 4.66 (.48)

26. Secondary Outcome: Severity of Depression in Caregivers
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 18 months.
Time Frame: 18-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 586 | 649 | 80
score on a scale | 4.34 (0.18) | 4.39 (0.17) | 4.19 (0.43)

27. Secondary Outcome: Severity of Depression in Caregivers (Common Baseline)
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the least squares mean of the baseline "treatment 0", which can be compared to the overall follow-up least square means to estimate treatment effects in each arm.
Time Frame: Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Common Baseline
Number analyzed (Participants) | 2174
score on a scale | 4.72 [4.52 to 4.95]

28. Secondary Outcome: Severity of Depression in Caregivers
Description: The severity of depression in caregivers as measured by the Patient Health Questionnaire (PHQ-8). PHQ-8 is an 8-item validated tool used to assess depressive symptoms in the caregiver using the Diagnostic and Statistical Manual IV (DSM-IV) criteria for major depression and is scored from 0-24 with scores >10 indicating moderate symptoms and scores >20 indicating severe depressive symptoms. The analyses are comparisons between each arm's average of its 3-month, 6-month, 12-month, and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents those average least squares means across all follow-up times for each arm.
Time Frame: Average of 3M, 6M, 12M, and 18M least square means
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1016 | 1014 | 144
score on a scale | 4.70 [4.47 to 4.94] | 4.42 [4.19 to 4.66] | 4.69 [4.17 to 5.22]
Statistical Analysis 1: Comparison: Health Systems-Based Dementia Care vs Community-Based Dementia Care; Test type: Superiority; p = 0.23, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = 0.28, 95% CI 2-sided [.01 to .54]
Statistical Analysis 2: Comparison: Health Systems-Based Dementia Care vs Usual Care; Test type: Superiority; p = .98, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons *three secondary outcomes; marginal difference of LS means = 0.01, 95% CI 2-sided [-.53 to .55]
Statistical Analysis 3: Comparison: Community-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.65, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = -0.27, 95% CI 2-sided [-0.81 to 0.27]

29. Secondary Outcome: Caregiver Self-Efficacy: 4-item Self-efficacy Scale
Description: Caregivers' ability to manage dementia-related problems and ability to access help is measured with a 4-item self-efficacy scale [range, 1 (strongly disagree) to 5 (strongly agree)] measuring the caregiver's self-efficacy for caring for the patient with dementia and for accessing help, including community resources. The scores for each of the 4 items are summed to produce an overall caregiver self-efficacy score ranging from 4-20 with higher scores indicating better caregiver self-efficacy. The analyses are comparisons between each arm's average of its 6-month and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1011 | 1011 | 143
score on a scale | 13.26 (.10) | 13.12 (.10) | 13.17 (.25)

30. Secondary Outcome: Caregiver Self-Efficacy: 4-item Self-efficacy Scale
Description: Caregivers' ability to manage dementia-related problems and ability to access help is measured with a 4-item self-efficacy scale [range, 1 (strongly disagree) to 5 (strongly agree)] measuring the caregiver's self-efficacy for caring for the patient with dementia and for accessing help, including community resources. The scores for each of the 4 items are summed to produce an overall caregiver self-efficacy score ranging from 4-20 with higher scores indicating better caregiver self-efficacy. The analyses are comparisons between each arm's average of its 6-month and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 6 months.
Time Frame: 6-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 793 | 812 | 112
score on a scale | 15.01 (0.10) | 15.00 (0.10) | 14.29 (0.32)

31. Secondary Outcome: Caregiver Self-Efficacy: 4-item Self-efficacy Scale
Description: Caregivers' ability to manage dementia-related problems and ability to access help is measured with a 4-item self-efficacy scale [range, 1 (strongly disagree) to 5 (strongly agree)] measuring the caregiver's self-efficacy for caring for the patient with dementia and for accessing help, including community resources. The scores for each of the 4 items are summed to produce an overall caregiver self-efficacy score ranging from 4-20 with higher scores indicating better caregiver self-efficacy. The analyses are comparisons between each arm's average of its 6-month and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the means of the raw outcome data for each arm at 18 months.
Time Frame: 18-month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 584 | 648 | 80
score on a scale | 15.09 (0.11) | 15.36 (0.11) | 14.66 (0.35)

32. Secondary Outcome: Caregiver Self-Efficacy: 4-item Self-efficacy Scale (Common Baseline)
Description: Caregivers' ability to manage dementia-related problems and ability to access help is measured with a 4-item self-efficacy scale [range, 1 (strongly disagree) to 5 (strongly agree)] measuring the caregiver's self-efficacy for caring for the patient with dementia and for accessing help, including community resources. The scores for each of the 4 items are summed to produce an overall caregiver self-efficacy score ranging from 4-20 with higher scores indicating better caregiver self-efficacy. The analyses are comparisons between each arm's average of its 6 and 18 months least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents the least squares mean of the baseline "treatment 0", which can be compared to the overall follow-up least square means to estimate treatment effects in each arm.
Time Frame: Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Common Baseline
Number analyzed (Participants) | 2172
score on a scale | 13.24 [13.10 to 13.39]

33. Secondary Outcome: Caregiver Self-Efficacy: 4-item Self-efficacy Scale
Description: Caregivers' ability to manage dementia-related problems and ability to access help is measured with a 4-item self-efficacy scale [range, 1 (strongly disagree) to 5 (strongly agree)] measuring the caregiver's self-efficacy for caring for the patient with dementia and for accessing help, including community resources. The scores for each of the 4 items are summed to produce an overall caregiver self-efficacy score ranging from 4-20 with higher scores indicating better caregiver self-efficacy. The analyses are comparisons between each arm's average of its 6-month and 18-month least squares means using a constrained longitudinal model that assigns all baseline data to a common "treatment 0." This entry presents those average least squares means across all follow-up times for each arm.
Time Frame: Average of 6M and 18M least square means
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1013 | 1015 | 144
score on a scale | 15.06 [14.89 to 15.23] | 15.22 [15.05 to 15.38] | 14.36 [13.95 to 14.78]
Statistical Analysis 1: Comparison: Health Systems-Based Dementia Care vs Community-Based Dementia Care; Test type: Superiority; p = 0.62, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = -0.16, 95% CI 2-sided [-0.37 to 0.06]
Statistical Analysis 2: Comparison: Health Systems-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.01, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = 0.70, 95% CI 2-sided [0.26 to 1.14]
Statistical Analysis 3: Comparison: Community-Based Dementia Care vs Usual Care; Test type: Superiority; p = 0.001, Mixed Models Analysis — Alpha = 0.05; Hochberg correction for three pairwise comparisons * three secondary outcomes; marginal difference of LS means = 0.85, 95% CI 2-sided [0.42 to 1.29]

34. Other Pre Specified Outcome: Cognition of Persons Living With Dementia
Description: Cognition as measured by the Montreal Cognitive Assessment (MoCA). MoCA is a validated widely used test of cognition that captures mild cognitive impairment as well as dementia. This will be collected at baseline by telephone and at the end of the study at 18 months to document disease progression.
  To reduce respondent burden and missing data, we will use a shortened 3-item form (a 0-12 point scale for evaluating memory, verbal fluency, and orientation only) for reporting study participant baseline characteristics and measuring the decline in cognition. Higher scores indicate less impairment. Participants who score 8 or higher on the shortened version will receive the full 22-item telephone MOCA to determine whether they have capacity to provide informed consent.
  This entry presents the means of the raw outcome data for each arm among PLWD who completed MoCA at baseline.
Time Frame: Baseline
Population: PLWD with completed MoCA at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 704 | 709 | 99
score on a scale | 6.2 (5.7) | 6.4 (6.0) | 5.9 (5.1)

35. Other Pre Specified Outcome: Cognition of Persons Living With Dementia (Missing Data)
Description: Cognition as measured by the Montreal Cognitive Assessment (MoCA). MoCA is a validated widely used test of cognition that captures mild cognitive impairment as well as dementia. This will be collected at baseline by telephone and at the end of the study to document disease progression.
  To reduce respondent burden and missing data, we will use a shortened 3-item form (a 0-12 point scale for evaluating memory, verbal fluency, and orientation only) for reporting study participant baseline characteristics and measuring the decline in cognition. Participants who score 8 or higher on the shortened version will receive the full 22-item telephone MOCA to determine whether they have capacity to provide informed consent.
  Report is among PLWD with missing MoCA at baseline.
Time Frame: Baseline
Population: PLWD with missing MoCA at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 312 | 307 | 45
Participants
  Hearing impairment | 115 | 121 | 15
  Participant refusal | 125 | 131 | 21
  Clinical decision | 52 | 39 | 7
  Partial data | 20 | 16 | 2

36. Other Pre Specified Outcome: Functional Status Measured by FAQ
Description: Functional status measured using the Functional Activities Questionnaire (FAQ). FAQ ranges from 0 to 30 with higher scores indicating more functional dependence. FAQ outcomes were collected at baseline and at 18 months. This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Population: PLWD with completed FAQ at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 999 | 997 | 143
score on a scale | 21.4 (7.5) | 21.3 (7.2) | 21.0 (8.0)

37. Other Pre Specified Outcome: Functional Status Measured by ADLs
Description: Functional status measured using Katz' Index of Independence in Activities of Daily Living (ADL) ranges from 0 to 6 with higher scores indicating more functional independence. Outcomes were collected at baseline and at 18 months. This entry presents the means of the raw outcome data for each arm at baseline.
Time Frame: Baseline
Population: PLWD with completed Katz at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
Number analyzed (Participants) | 1013 | 1010 | 144
score on a scale | 4.4 (1.9) | 4.5 (1.8) | 4.5 (1.8)

38. Other Pre Specified Outcome: Goal Attainment
Description: Asks patients & caregivers to select their most important goal and assesses their progress towards meeting it as a result of one of the study's intervention. Goal attainment, defined as whether a person's individual goals are achieved as a result of the study intervention, will be measured using a 5-point goal attainment scale (GAS). GAS describes the person's expected level of goal achievement over a specified timeframe, ranging from much worse than expected (scored as -2) to much better than expected (scored as +2). Scales are dynamically set according to a person's needs, while measurement of attainment is standardized. The outcome will be a least squares marginal mean based on follow-up measurements at 6 and 18 months.
Time Frame: 18 months
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Number of Persons With Dementia That Die Over the Course of the Study
Description: Mortality of persons with dementia as measured by interviews with caregivers at 3, 6, 12, and 18 months. Data will be verified using the Center for Medicare and Medicaid Services at 18 months. For participants who did not complete the 18-month interview, vital status will be investigated using the electronic health records (EHR).
Time Frame: 18 months
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Time Spent at Home
Description: Time spent at home is defined as [number of days since randomization - (number of inpatient days spent at an acute care hospital, inpatient rehabilitation facility, skill nursing facility, long-term care facility, or inpatient hospice unit)/Number of days since randomization].
Time Frame: 18 months
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Caregiver Rating of Dementia Care Quality
Description: Caregiver Rating of Dementia Care Quality is a composite instrument of 10 items (with yes or no responses) from the Assessing Care of Vulnerable Elders (ACOVE), Physician Consortium for Performance Improvement (PCPI) and the American Academy of Neurology (AAN) quality measures. The outcome is a count of the number of yes responses (range 0-10, higher counts indicate greater caregiver rating of satisfaction of dementia care quality).
Time Frame: 12 months
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Caregiver Assessment of Dementia Care
Description: Caregiver's satisfaction with the dementia care program is measured using a 11-item questionnaire, modified from the University of California Los Angeles' Alzheimer's and Dementia Care program, with ranges from 11 to 55 (higher scores indicate greater caregiver satisfaction with the dementia care program). The questionnaire will be administered at 3, 12 and 18 months.
Time Frame: 18 months
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Dementia Burden (Caregiver)
Description: Dementia Burden Scale-Caregiver (DBS-CG) is a composite of the NPI-Q Distress, MCSI, and PHQ-8 scales with items transformed linearly to be on a 0-100 possible range and then averaged with higher scores indicating higher caregiver burden. The minimal clinically important difference (MCID) for the DBS-CG is 5 points. The outcome will be a least squares marginal mean based on follow-up measurements at 3, 6, 12 and 18 months.
Time Frame: 18 months
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Clinical Benefit
Description: Clinical benefit is a binary measure of patient symptoms using the NPI-Q severity scale (the only patient outcome anticipated to benefit from the program) and caregiver symptoms using the DBS-CG scale. Benefit on the NPI-Q severity scale is defined as having a 1-year score of less than or equal to 6 (the lowest tertile of symptoms) or improving by at least 3 points, the MCID. DBS-CG benefit is defined as having a 1-year score of less than or equal to 18.8 (the lowest tertile of symptoms) or improving by at least 5 points, the MCID. Defining benefit in this manner captures both preventive (those who have few symptoms at baseline and do not deteriorate) and therapeutic (those who improve) benefit from the program. The outcome will be an overall odds ratio based on follow-up measurements at 3, 6, 12 and 18 months.
Time Frame: 18 months
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Quality of Life of People With Dementia: QOL-AD
Description: Quality of life as measured by the Quality of Life in Alzheimer's Disease (QOL-AD). The QOL-AD is a 13-item instrument scored 4-52 (higher scores indicate better quality of life) that can be administered to persons with dementia and caregivers. It has demonstrated sensitivity to psychosocial intervention correlates with health-utility measures, is widely translated and used internationally and can be used by people with Mini-Mental State Exam (MMSE) scores as low as three. The outcome will be measured at 18 months.
Time Frame: 18 months
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Positive Aspects of Family Caregiving
Description: The positive aspects of family caregiving as measured by the Positive Aspects of Family Caregiving Questionnaire, which is an 11-item tool to assess favorable aspects of caregiving experiences, and is scored from 0 to 44 (most positive) with higher scores indicating a more positive mental and affective state related to the caregiver's experience. The outcome will be measured at 6 months.
Time Frame: 6 months
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Inpatient Days Spent at an Acute Care Hospital
Description: Inpatient Days Spent at an Acute Care Hospital is defined as the number of days an individual is admitted to an acute care hospital. This outcome will be attained using data from the Centers for Medicare and Medicaid Services (CMS).
Time Frame: 18 months
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Inpatient Days Spent at an Inpatient Rehabilitation Facility
Description: Inpatient Days Spent at an Inpatient Rehabilitation Facility is defined as the number of days an individual is admitted to an inpatient rehabilitation facility. This outcome will be attained using data from CMS.
Time Frame: 18 months
Reporting Status: Not Posted

49. Other Pre Specified Outcome: Inpatient Days Spent at a Skilled Nursing Facility
Description: Inpatient Days Spent at a Skilled Nursing Facility is defined as the number of days an individual is admitted to a Skilled Nursing Facility. This outcome will be attained using data from CMS.
Time Frame: 18 months
Reporting Status: Not Posted

50. Other Pre Specified Outcome: Inpatient Days Spent at a Long-term Care Facility
Description: Inpatient Days Spent at a Long-term Care Facility is defined as the number of days an individual is admitted to a Long-term Care Facility. This outcome will be attained using data from CMS.
Time Frame: 18 months
Reporting Status: Not Posted

51. Other Pre Specified Outcome: Placement in Long-term Care Facility
Description: Placement in a Long-term Care Facility is defined by (1) observed placement in a long-term care facility, or (2) the time (days) from enrollment to when individual is admitted to a Long-term Care Facility. This outcome will be attained using data from CMS.
Time Frame: 18 months
Reporting Status: Not Posted

52. Other Pre Specified Outcome: Days Spent Receiving Hospice Benefit
Description: Days Spent Receiving Hospice Benefit is defined as the number of days an individual is receiving hospice care regardless of location. This outcome will be attained using data from CMS.
Time Frame: 18 months
Reporting Status: Not Posted

53. Other Pre Specified Outcome: Physician Assessment of Dementia Care at 18 Months
Description: The level of physician satisfaction with dementia care programs as measured by the Physician Assessment of Dementia Care (PADC). The PADC is an 5-item questionnaire modified from UCLA's Alzheimer's and Dementia Care program. Each item will be examined individually (with the range of each item differing). The questionnaire will be administered at 18 months, when the provider's first enrolled patient completes the study. All providers with at least one enrolled patient in the study will be surveyed.
Time Frame: 18 months
Reporting Status: Not Posted

54. Other Pre Specified Outcome: Cost-Effectiveness Relative to Severity of Dementia-related Behavioral Symptoms
Description: The cost-effectiveness of the interventions compared to usual care is the ratio of incremental net costs to incremental effects of the NPI-Q-Severity. Thus, the ratio will be the net costs per unit change in NPI-Q-Severity. Costs will be taken from the perspective of Medicare. The net costs of the interventions are the costs of training for and doing the intervention less the cost offsets of reduced medical care and caregiving, if any, they bring about. The intervention costs, primarily labor, will be collected at the sites.
Time Frame: 18 months
Reporting Status: Not Posted

55. Other Pre Specified Outcome: Cost-Effectiveness Relative to Caregiver Distress
Description: The cost-effectiveness of the interventions compared to usual care is the ratio of incremental net costs to incremental effects of the Modified Caregiver Strain Index (MCSI). Thus, the ratio will be the net costs per unit change in MCSI. Costs will be taken from the perspective of Medicare. The net costs of the interventions are the costs of training for and doing the intervention less the cost offsets of reduced medical care and caregiving, if any, they bring about. The intervention costs, primarily labor, will be collected at the sites.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Enrollment through death, withdrawal, or 18 months of follow-up
Description: Other (Not Including Serious) Adverse Events were not monitored/assessed in the study.
  Deaths and overnight hospitalizations of Persons Living with Dementia (PLWD) were ascertained by caregiver report. Caregiver Serious Adverse Events were not collected in the study.
Arm/Group | Health Systems-Based Dementia Care | Community-Based Dementia Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 254/1016 | 223/1016 | 37/144
Serious Adverse Events (participants affected / at risk) | 528/1016 | 533/1016 | 70/144
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Systems-Based Dementia Care (N=1016) | Community-Based Dementia Care (N=1016) | Usual Care (N=144)
Allergic (Immune system disorders) | 2 (2) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 21 (26) | 26 (32) | 3 (3)
Cardiopulmonary (Cardiac disorders) | 64 (86) | 60 (78) | 9 (14)
Cardiopulmonary (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 31 (41) | 2 (2)
Endocrine or Metabolic (Endocrine disorders) | 10 (14) | 3 (3) | 1 (1)
Falls or fractures (Musculoskeletal and connective tissue disorders) | 98 (118) | 82 (101) | 8 (9)
Gastroenterologic (Gastrointestinal disorders) | 26 (30) | 35 (43) | 8 (8)
Hematologic (Hepatobiliary disorders) | 2 (2) | 5 (7) | 2 (2)
Infection (Infections and infestations) | 88 (110) | 72 (108) | 13 (18)
Neurologic (Nervous system disorders) | 63 (79) | 76 (86) | 12 (14)
Neuropsychiatric complications of dementia (Psychiatric disorders) | 18 (20) | 16 (19) | 1 (1)
Oncologic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 6 (8) | 0 (0)
Renal or electrolytes (Renal and urinary disorders) | 18 (25) | 26 (38) | 4 (4)
Surgical procedure other than fracture repair (Surgical and medical procedures) | 17 (20) | 16 (16) | 4 (4)
Unknown/Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Unknown/Other (Cardiac disorders) | 4 (8) | 6 (7) | 1 (2)
Unknown/Other (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Unknown/Other (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Unknown/Other (General disorders) | 24 (36) | 31 (45) | 0 (0)
Unknown/Other (Infections and infestations) | 3 (4) | 12 (12) | 0 (0)
Unknown/Other (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Unknown/Other (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 0 (0)
Unknown/Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Unknown/Other (Nervous system disorders) | 5 (5) | 4 (5) | 0 (0)
Unknown/Other (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Unknown/Other (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Unknown/Other (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Unknown/Other (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Unknown/Other (Surgical and medical procedures) | 3 (3) | 2 (2) | 0 (0)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (14) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT03786471/Prot_002.pdf
  • Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03786471/SAP_000.pdf
  • Informed Consent Form (2023-08-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03786471/ICF_001.pdf